CLINICAL TRIAL: NCT04375527
Title: A Phase 2 Study of Combination Treatment of Binimetinib and Nivolumab for Advanced V600BRAF Wildtype Melanoma with Innate Anti-PD-1 Resistance
Brief Title: Binimetinib and Nivolumab for the Treatment of Locally Advanced Unresectable or Metastatic BRAF V600 Wildtype Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Array BioPharma (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-002060; NCI-2020-02590 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC V8; Clinical Stage IV Cutaneous Melanoma AJCC V8; Locally Advanced Cutaneous Melanoma; Metastatic Cutaneous Melanoma; Pathologic Stage III Cutaneous Melanoma AJCC V8; Pathologic Stage IIIA Cutaneous Melanoma AJCC V8; Pathologic Stage IIIB Cutaneous Melanoma AJCC V8; Pathologic Stage IIIC Cutaneous Melanoma AJCC V8; Pathologic Stage IIID Cutaneous Melanoma AJCC V8; Pathologic Stage IV Cutaneous Melanoma AJCC V8; Unresectable Cutaneous Melanoma
MeSH Terms: conditions — Melanoma | interventions — binimetinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (binimetinib, nivolumab) (Experimental): Patients receive binimetinib PO BID on days 1-28 and nivolumab IV over 30 minutes on day 1. Treatment repeats every 4 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib; Biological: Nivolumab; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY-162; ARRY-438162; MEK162; Mektovi
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well binimetinib and nivolumab work in treating patients with BRAF V600 wildtype melanoma that has spread to nearby tissues or lymph nodes and cannot be removed by surgery (locally advanced unresectable) or has spread to other places in the body (metastatic). Binimetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving binimetinib and nivolumab together may work better in treating patients with melanoma compared to nivolumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Objective response rate (ORR), which is defined as the proportion of response-evaluable participants either with a confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, as determined by the investigator assessment, at best overall response.

SECONDARY OBJECTIVE:

I. Progression-free survival (PFS), clinical benefit rate (CR + PR + stable disease [SD] among response-evaluable participants, per RECIST 1.1), overall survival (OS) and duration of response (DOR).

EXPLORATORY OBJECTIVE:

I. Evaluation of histologic evidence of response (p-ERK reduction in residual tumor cells and CD8 T cell or tumor infiltrating lymphocytes or tumor infiltrating lymphocyte [TIL] infiltration induced by combination treatment) using pretreatment and early on-treatment tumor biopsies.

OUTLINE:

Patients receive binimetinib orally (PO) twice daily (BID) on days 1-28 and nivolumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 4 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 1 year, then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Histologically confirmed locally advanced/unresectable or metastatic cutaneous melanoma
* Measurable disease per RECIST version (v.) 1.1 criteria using imaging scans, OR peripheral lesions that can be adequately documented with a picture and a ruler even if they do not meet RECIST criteria
* Patient must have failed prior alphaPD-1 or alphaPD-1 + alphaCTLA-4 therapy in the metastatic setting
* V600BRAF wildtype tumor status confirmed by Clinical Laboratory Improvement Act (CLIA) approved lab
* Hemoglobin >= 8.0 g/dL
* Whole blood cell count (WBC) >= 2,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 75,000/mm^3
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x institutional upper limit of normal (ULN), (=< 5.0 x ULN in those with hepatic metastases)
* Bilirubin =< 1.5 x ULN; for subjects with documented/suspected Gilbert's disease, bilirubin =< 3 x ULN
* Albumin >= 2.5 g/dl
* Serum creatinine =< 2.0 x upper limit of normal (ULN)
* Left ventricular ejection fraction (LVEF) >= 50% assessed by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan completed =< 180 days (6 months) before initiation of protocol treatment
* Patients must be willing to submit blood and tissue specimens for translational medicine studies
* Patients must have a site of disease amenable to biopsy and be a candidate for biopsy
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) at screening and within 24 hours prior to the start of study drug
* Women of childbearing potential (WOCBP) must be willing to use either two adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy, or to abstain from heterosexual activity (complete abstinence) throughout the study, starting with visit 1 through 5 months after the last dose of study therapy. Approved contraceptive methods include, for example, intrauterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, female condoms with spermicide, or oral contraceptives. Spermicides alone are not an acceptable method of contraception. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Male patients must agree to use an adequate method of contraception, or to abstain from heterosexual activity (complete abstinence) starting with the first dose of study drug through 5 months after the last dose of study therapy

Exclusion Criteria:

* Contraindications to tumor biopsy (coagulopathy, known history of keloid formation, etc.)
* Women who are pregnant or breastfeeding
* Prior therapy with a MEK inhibitor (e.g., binimetinib, trametinib, cobimetinib)
* Known hypersensitivity or contraindication to any component of binimetinib or its excipients
* Inability to swallow and retain study drug
* Patients who have received prior lines of systemic therapy in the advanced/metastatic setting (not including, neoadjuvant, adjuvant, or maintenance therapy)
* Received anticancer therapy including chemotherapy, immunotherapy, or antineoplastic biologic therapy (e.g., erlotinib, cetuximab, bevacizumab etc.), within 14 days prior to start of study treatment or exposure to any investigational drug within 7 days prior to screening visit or for which 5 half-lives have not elapsed
* Participants who have undergone major surgery (e.g., in-patient procedures) =< 6 weeks prior to start of study treatment or who have not recovered from side effects of such procedure
* Participants who have had radiotherapy =< 14 days prior to start of study treatment or who have not recovered from side effects of such procedure. Note: Palliative radiation therapy must be complete 7 days prior to the first dose of study treatment
* Participants who have not recovered to =< grade 1 from toxic effects of prior therapy before starting study treatment

  * Note: Stable chronic conditions (=< grade 2) that are not expected to resolve (such as neuropathy, myalgia, alopecia, prior therapy-related endocrinopathies) are exceptions and may enroll
* Uncontrolled or symptomatic brain metastases or leptomeningeal carcinomatosis that are not stable, require steroids, are potentially life-threatening or have required radiation within 28 days prior to starting study drug. Note: Patients with previously treated brain metastases may participate provided they are stable (e.g., without evidence of progression by radiographic imaging for at least 28 days before the first dose of study treatment and neurologic symptoms have returned to baseline), and have no evidence of new or enlarging brain metastases or central nervous system (CNS) edema, and does not require steroids at least 7 days before the first dose of study treatment
* Subjects with active, known, or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

  * Myocardial infarction (MI) or stroke/transient ischemic attack (TIA) within the 6 months prior to consent
  * Uncontrolled angina within the 3 months prior to consent
  * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, torsades de pointes, or poorly controlled atrial fibrillation)
  * Corrected QT (QTc) prolongation > 480 msec
  * History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association [NYHA] functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, poorly controlled deep venous thrombosis, etc)
  * Cardiovascular disease-related requirement for daily supplemental oxygen
  * History of two or more myocardial infarctions OR two or more coronary revascularization procedures
  * Subjects with history of myocarditis, regardless of etiology
  * History of thromboembolic or cerebrovascular events =< 12 weeks prior to the first dose of study treatment. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or sub-massive) deep vein thrombosis or pulmonary emboli

    * Note: Patients with either deep vein thrombosis or pulmonary emboli that does not result in hemodynamic instability are allowed to enroll as long as they are on a stable dose of anticoagulants for at least 4 weeks
    * Note: Patients with thromboembolic events related to indwelling catheters or other procedures may be enrolled
* A confirmed history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent
* Participants with a condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent)
* Subjects receiving any other investigational or standard antineoplastic agents
* Patients with severe grade 3-4 toxicities due to anti-PD-1 monotherapy during first line. Toxicities due to combination PD-1/CTLA-4 blockade will not be exclusionary
* Inability to give informed consent
* History of malignancies except cured basal cell carcinoma, cutaneous squamous cell carcinoma, melanoma in situ, superficial bladder cancer or carcinoma in situ of the cervix; for other malignancies, must be documented to be free of cancer for >= 2 years. All other cases can be considered on a case by case basis at the discretion of the principal investigator
* Any condition that might interfere with the subject's participation in the study, safety, or in the evaluation of the study results
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study
* Active or prior documented inflammatory bowel disease
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids or has current ILD/pneumonitis or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Impairment of gastrointestinal function or disease which may significantly alter the absorption of study drug (e.g., active ulcerative disease, uncontrolled vomiting or diarrhea, malabsorption syndrome, small bowel resection with decreased intestinal absorption), or recent (=< 3 months) history of a partial or complete bowel obstruction, or other conditions that will interfere significantly with the absorption of oral drugs
* Concurrent neuromuscular disorder that is associated with elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* History or current evidence of retinal venous occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of retinal degenerative disease
* Prisoners or subjects who are involuntarily incarcerated

  * Note: under certain specific circumstances a person who has been imprisoned may be included or permitted to continue as a subject
  * Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Up to 26 months
  Will be defined as the total number of patients with confirmed responses of either complete response or partial response divided by the total number of subjects in the enrolled population per Response Evaluation Criteria in Solid Tumors 1.1 by investigator assessment. Will be calculated along with the corresponding exact one-sided 95% Clopper-Pearson confidence interval.

SECONDARY OUTCOMES:
Progression-free survival | From first dose of study drug to the date of progressive disease first documented disease progression or death due to any cause by investigator assessment, or the start of secondary antitumor therapy, whichever occurs first, assessed up to 26 months
  Will be assessed per Response Evaluation Criteria in Solid Tumors 1.1. Will be summarized using the Kaplan Meier method. Will be summarized descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum). Figures showing the Kaplan-Meier estimates will also be presented.
Clinical benefit rate | Up to 26 months
  Will be defined as the proportion of response-evaluable participants who have achieved a confirmed complete response, partial response, and stable disease per Response Evaluation Criteria in Solid Tumors 1.1, as determined by the investigator assessment. Clinical benefit rate and the individual rates for complete response/partial response/stable disease will be summarized with the frequency count and the percentage of subjects in each category along with a 2-sided 95% exact confidence interval.
Overall survival | From first dose of study drug and death due to any cause, assessed up to 26 months
  Will be summarized using the Kaplan Meier method. The Kaplan Meier estimates for the 1 year OS rates and the 2-sided 95% confidence interval of the rates using the Greenwood's formula will be reported. Will be summarized descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum). Figures showing the Kaplan-Meier estimates will also be presented.
Duration of response | From the time measurement criteria is met for complete response/partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 26 months
  Will be summarized using the Kaplan Meier method. Will be summarized descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum). Figures showing the Kaplan-Meier estimates will also be presented.

OTHER OUTCOMES:
Pharmacodynamic marker analysis | Up to disease progression, assessed up to 26 months
  Will use purely descriptive analysis to assess biomarkers (PDL1 status at baseline, baseline mutational load, presence of tumor infiltrating lymphocytes, hormone receptor status, T-cell receptor repertoire in tumor infiltrating lymphocytes and peripheral blood mononuclear cells). They will be further related to individual subject tumor responses.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Lo, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States